CLINICAL TRIAL: NCT01132365
Title: Knee Arthroplasty Registry a. Function and Survival Stratified by BMI b. Return of Quadriceps Strength After Primary TKA
Brief Title: Knee Arthroplasty Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heekin Orthopedic Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry); Stryker Orthopaedics (Industry); Restor3D (Industry)
Responsible Party: Principal Investigator, R. David Heekin, MD, R. David Heekin, M.D., Heekin Orthopedic Research Institute
Other Study IDs: 05-05-02
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis, Knee
Keywords: knee arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- knee arthroplasty
  Interventions: Device: any knee joint arthroplasty device

INTERVENTIONS:
Device: any knee joint arthroplasty device — Cohort consist of all consented patients receiving knee arthroplasty
  Other Names: Total Knee Arthoplasty; Unicondylar Knee arthroplasty; Revision Knee Arthroplasty

SUMMARY:
Objective

Describe the clinical and demographic characteristics of patients who undergo knee arthroplasty and document post operative outcomes.

Examine the relationship between processes of care, hospital and surgeon associated outcomes.

Provide expanded data to characterize existing and evolving practice patterns, delivery of care, and resource utilization in the management of knee arthroplasty patients.

Analyze and design ancillary studies to address unanswered questions.

Disseminate findings through publication in peer-reviewed scientific journals.

DETAILED DESCRIPTION:
Population: All male and non-pregnant females undergoing knee arthroplasty.

Study Design: Prospective, consecutive series on an unlimited number of patients.

Data Collection

Clinic Data:

Patient Demographics- age, weight, height, gender, affected side, co-morbidities, current medications, and contact information Knee Society Score SF-12 Evaluation of radiographs- AP, ML, and merchant view Preop lab results

Surgical Data:

Surgical approach ASA level Size of implants, catalog and lot numbers Time of surgery Estimated blood loss (ml) Length of incision (cm) Intraoperative ROM Any peculiar findings (i.e. heterotopic bone, large osteophytes, etc.) Preop lab results

Postoperative Data Sf-12 Modified Knee Society Score Quad strength testing Evaluation of radiographs, AP, ML, and merchant view

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a male or non-pregnant female over the age of 21.
2. Patient requires a knee arthroplasty, revision knee arthroplasty, or unicondylar knee arthroplasty
3. Patient has signed and dated an IRB approved consent form.
4. Patient is able and willing to participate in the study according to the protocol for the full length of expected term of follow-up, and to follow their physician's directions.
5. Patient has failed to respond to conservative treatment modalities.

Exclusion Criteria:

1. Patient's bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
2. Patient is a prisoner.

Ages: 21 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male and non-pregnant females undergoing knee arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 7793 (Estimated)
Dates: Start 2005-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | 2 weeks, 6 weeks, 3 months, 6 months, 1, 2, 5, 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Heekin, MD, Principal Investigator — Heekin Orthopedic Specialists
Locations (1):
- Heekin Orthopedic Specialists, Jacksonville, Florida, United States